CLINICAL TRIAL: NCT03956745
Title: Proteomic and Transcriptomic Biomarkers of Circadian Timing
Brief Title: Biomarkers for Circadian Timing in Healthy Adults
Status: Terminated | Type: Observational
Why Stopped: Grant funding supporting the study ended.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Stanford University (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jeanne Duffy, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2019-P-001247
Record Dates: First submitted 2019-04-23; First posted 2019-05-21 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Sleep Wake Disorders; Sleep Disorders, Circadian Rhythm; Sleep Disorders, Intrinsic; Advanced Sleep Phase Syndrome (ASPS); Advanced Sleep Phase Syndrome; Advanced Sleep Phase; Delayed Sleep Phase; Delayed Sleep Phase Syndrome; Non-24 Hour Sleep-Wake Disorder; Irregular Sleep-Wake Syndrome; Shift-Work Sleep Disorder; Shift Work Type Circadian Rhythm Sleep Disorder; Delayed Phase Sleep Syndrome
Keywords: Sleep; Aging; Circadian Rhythms; Circadian Rhythm Disorders
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Disorders, Circadian Rhythm; Sleep Disorders, Intrinsic; Chronobiology Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A genetic blood sample will be collected from each participant. Candidate circadian or sleep genes will be directly sequenced in order to identify polymorphisms or mutations that associate with circadian or sleep phenotypes. Researchers may also conduct genome wide analysis on the DNA sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: sleep-wake timing — Study participants will have one inverted day when they are scheduled to sleep ~12h opposite their usual sleep time.
Behavioral: constant routine — Study participants will spend ~28-50 hours awake, inactive, sitting in bed, in constant lighting and temperature.

SUMMARY:
Study investigators want to learn more about the underlying biological clock and to see if the timing of that clock can be estimated from a single blood sample.

DETAILED DESCRIPTION:
There is an urgent need for a practical way to assess circadian timing accurately in both general and sleep medicine. The study is designed to assess the levels of different biomarkers in the blood taken from frequent samples across three separate sleep-wake conditions - Conventional/Normal sleep-wake conditions (baseline), extended wake/acute sleep deprivation (constant routine), and during irregular sleep-wake conditions (inverted day). Participants will be asked to complete medical, psychological, and sleep-wake evaluations prior to the study. Upon completion of screening, if eligible, participants will stay 7 consecutive days and nights in the sleep research laboratory within the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with conventional and regular sleep-wake timing
* Non-smokers
* Able to spend 7 consecutive days/nights in the laboratory
* Willing to abstain from use of caffeine, nicotine, and alcohol during pre-study and study periods

Exclusion Criteria:

* History of neurological or psychiatric disorder
* History of sleep disorder or regular use of sleep-promoting medication
* Current prescription, herbal, or over-the-counter medication use
* Traveling across 2 or more time zones within the past 3 months
* Donating blood within the past 8 weeks
* Worked night or rotating shiftwork within the past 3 years
* Hearing impairment
* Drug or Alcohol dependency
* Pregnant, intending to become pregnant, or recently pregnant (last 6 months)
* Breastfeeding within the past 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be recruited from the surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Circadian Phase Timing by BodyTime Assay - Baseline Segment | Baseline Segment (Study day 3)
  Circadian phase will be predicted by the BodyTime assay during the baseline segment (study day 3) and will be compared to conventional phase assessment methods.
Circadian Phase Timing by BodyTime Assay - Constant Routine | During Constant Routine (Study days 4-5)
  Circadian phase will be predicted by the BodyTime assay during the Constant Routine (study days 4-5) and will be compared to conventional phase assessment methods.
Circadian Phase Timing by BodyTime Assay - Inverted Day | Inverted Day (Study days 6-7)
  Circadian phase will be predicted by the BodyTime assay during the Inverted Day (study days 6-7) and will be compared to conventional phase assessment methods.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne F Duffy, MBA, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States